CLINICAL TRIAL: NCT04364880
Title: Neuropsychobiology of Brain Theta-burst Stimulation: A Mind-body Interface for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuan-Pin, China Medical University Hospital, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NHRI-EX101-10144NI
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Depression; Treatment
Keywords: depression; transcranial magnetic stimulation; theta-burst stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theta-burst stimulation (TBS) (Experimental): Theta-burst stimulation (TBS) is a novel repetitive transcranial magnetic stimulation (rTMS)
  Interventions: Device: TBS
- Sham controlled intervention (Sham Comparator): The sham-TBS coil produced a similar sound without a magnetic pulse.
  Interventions: Device: Sham

INTERVENTIONS:
Device: TBS — Theta-burst stimulation (TBS) is a novel repetitive transcranial magnetic stimulation (rTMS)
  Arms: Theta-burst stimulation (TBS)
Device: Sham — The sham-TBS coil produced a similar sound without a magnetic pulse.
  Arms: Sham controlled intervention

SUMMARY:
This is a sham-controlled, randomized trial for patients with MDD to identify the effects of TBS on depressive symptomatology, brain function, and peripheral biomarkers in MDD patients.

DETAILED DESCRIPTION:
This is a sham-controlled, randomized trial for patients with MDD to identify the effects of TBS on depressive symptomatology, brain function (e.g. functional MRI, PET, and qEEG), peripheral biomarkers (e.g. candidate genetic expression, neuroendocrine, inflammation, and neurotransmissions) in MDD patients.

ELIGIBILITY:
Inclusion Criteria:

* The diagnostic criteria of DSM-IV for MDD
* The range of the age from 18 to 70-year-old
* Physically healthy on medical history, physical examination, and laboratory parameters within normal limits
* Competent for a full explanation of the study and written informed consent is obtained.

Exclusion Criteria:

* Having other current Axis I disorders (except nicotine dependence), patients with psychotic disorders, bipolar disorders, organic mental disorders, and a prevailing strong suicidal risk were excluded
* Pregnant
* History or family history of seizure disorder
* Known neurological disorders or evidence of central nervous system disease based on baseline complete neurological examination, electroencephalography, and magnetic resonance imaging of the brain
* Having ferromagnetic material in the body or close to the head (implanted pacemaker or medication pump, metal plate in skull, or metal objects in the eye or skull)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAMD) | From Weeks 0 to 24
  The Hamilton Depression scale sum score (HAMD21)
  * Not depressed: 0-7
  * Mild: 8-13
  * Moderate: 14-18
  * Severe: 19-22
  * Very severe: >23

SECONDARY OUTCOMES:
Response rate | From Weeks 0 to 24
  The decreasing level of the Hamilton Rating Scale for Depression from 0% to 50% compared to the sham group.
Remission rate | From Weeks 0 to 24
  The higher scores on the Hamilton Rating Scale for Depression down to 8 points would be considered remission.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Pin Su, MD PhD, Principal Investigator — China Medical University Hospital